CLINICAL TRIAL: NCT03388905
Title: Role of the Wearable Cardioverter Defibrillator in Tachycardia Induced Cardiomyopathy. A Prospective Study
Brief Title: Role of the Wearable Cardioverter Defibrillator in Tachycardia Induced Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ilan Goldenberg, MD, Professor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TICMP
Record Dates: First submitted 2017-12-03; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Tachycardia-induced Cardiomyopathy
Keywords: LifeVest wearable; cardioverter defibrillator; LVEF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Wearable Cardioverter Defibrillator group (Experimental)
  Interventions: Device: Life Vest Wearable defibrilator

INTERVENTIONS:
Device: Life Vest Wearable defibrilator — The LifeVest is a cardioverter defibrillator worn by a patient at risk for sudden cardiac arrest (SCA). It monitors the patient's heart continuously and, if the patient goes into a life-threatening arrhythmia, can deliver a shock treatment to restore the patient's heart to normal rhythm.

SUMMARY:
The purpose of this current study is to prospectively enroll consecutive patients hospitalized with newly diagnosed severe left ventricular dysfunction (LVEF ≤ 35%) for which the likely etiology is uncontrolled atrial fibrillation or high burden of ventricular ectopy. Patients completing their established in-hospital treatment plan with rate or rhythm control, will be discharged with a WCD following informed consent and detailed counseling by healthcare personnel for a time-period of up to 3 months until reassessment of LVEF and the need for ICD implantation.

DETAILED DESCRIPTION:
TachycardiaInduced Cardiomyopathy (TICMP) refers to impairment in left ventricular function secondary to chronic tachycardia, which is partially or completely reversible once the tachyarrhythmia is controlled. Tachycardia-induced cardiomyopathy has been shown to occur both in experimental models and in patients with incessant tachyarrhythmia (mostly commonly uncontrolled atrial fibrillation). Control of ventricular rate or rhythm by means of cardio-version, negative chronotropic agents, anti-arrhythmic medication and surgical or catheter-based ablation, resulted in significant improvement of systolic function. However, until a possible improvement in left ventricular ejection fraction (LVEF), patients with TICMP with severely depressed systolic function may remain at a high-risk for life-threatening ventricular arrhythmias and sudden cardiac death. While implantable cardioverter defibrillators (ICD) are indicated in patients who fail to improve their left ventricular ejection fraction (LVEF), currently there is no protection from sudden cardiac death (SCD) in patients with TICMP during the high-risk time period from hospital discharge until reassessment of cardiac function and the need for ICD implantation. In this population, the Life Vest wearable cardioverter defibrillator (WCD) may be an appropriate treatment option, providing protection from SCD through timely termination of life-threatening ventricular arrhythmias until stabilization of LVEF. In addition, the monitoring capabilities of the WCD may facilitate remote assessment heart rate control with appropriate titration of medical therapy and evaluation of recurrence of tachyarrhythmias following discharge from hospitalization. Accordingly, the proposed study is the first to prospectively evaluate the benefit of the WCD as an early management strategy in patients with TICMP.

There is no available clinical research data to date on the study device used in TICMP.

This proposed trial is a multicenter single armed prospective study. Thirty patients with newly diagnosed severe LV dysfunction due to uncontrolled tachyarrhythmia will be enrolled following their completion of established in-hospital treatment plan with rate or rhythm control.

Enrolled patients will be discharged with a WCD for a time-period of 3 months. All patients will provide signed informed consent, and detailed counseling by healthcare personnel for a time-period of up to 3 months until reassessment of LVEF and the need for ICD implantation.

The enrollment duration is expected to last 12 months and follow up of additional 12 months from patient inclusion will be performed. An estimation recruitment rate of 1-2 patients per month per center is reasonable based on our preliminary data (see section 6.1). Therefore, it is likely to end up patient's recruitment 10 months following the enrollment phase initiation.

During follow up, patients will be contacted at (1) end of WCD use (2) 3 month and (3) 12 months post enrollment.

Total expected duration of study termination is 24 months from the time first patient was enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed left ventricular dysfunction (LVEF ≤ 35% following cardioversion or rate stabilization) with either of the following:

  * Newly diagnosed atrial fibrillation
  * High burden of premature ventricular contractions (PVCs) (15% of total beats on 24-hour ambulatory Holter recording with a rapid ventricular response > 100 beats per minute prior to initiation of medical therapy) and no other likely heart failure (HF) etiology
* Appropriate management during hospitalization with cardioversion and rhythm control (preferable) or rate control (if cardioversion is contraindicated due to a left atrial thrombus or is not successful)

Exclusion Criteria:

* HF likely due to an etiology other than tachyarrhythmia (ischemic etiology, myocarditis, hypertrophic or dilated cardiomyopathy, etc.)
* Unstable clinical condition, life threatening arrhythmia or an established indication for ICD/CRT-D implantation during the index hospitalization
* Patients with ICD/CRT-D or established (> 3 months) heart failure
* Cognitive impairment or unable to utilize WCD appropriately
* Patient has a chest circumference at the level of the xiphoid process either less than 26 inches or greater than 56 inches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular recovery following WCD use. | 3 months
  Left ventricular recovery following WCD use.

SECONDARY OUTCOMES:
Recurrence of atrial tachyarrhythmias | 12 months
  Recurrence of atrial tachyarrhythmias
Recurrence of ventricular tachyarrhythmias | 12 months
  Recurrence of ventricular tachyarrhythmias
Appropriate shocks by WCD | 3 months
  Occurrence of appropriate shocks as recorded by WCD (number of Shocks delivered during the follow up period)
Inappropriate shocks by WCD | 3 months
  Occurrence of Inappropriate shocks as recorded by WCD (number of Inappropriate Shocks delivered during the follow up period)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No